CLINICAL TRIAL: NCT03185585
Title: Development and Validation of a Comprehensive Older Adult Screening Tool (COAST)
Brief Title: Validation of a Comprehensive Older Adult Screening Tool (COAST)
Acronym: COAST
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201701083
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Community-dwelling Older Adults
Keywords: Nutritional screenings
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults 60 yrs and older: Participants will be asked to take the full MNA and COAST tools, separately .They will take a hand grip strength test to evaluate their functional status and five times Sit to Stand test as part of the COAST screening tool. Moreover, their weight, height, mid-arm circumference and calf circumference, will be measured as part of the MNA screening tool.
  Interventions: Other: Mini Nutrition Assessment (MNA® ); Other: Comprehensive Older Adult Screening Tool (COAST)

INTERVENTIONS:
Other: Mini Nutrition Assessment (MNA® ) — MNA® is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition.
Other: Comprehensive Older Adult Screening Tool (COAST) — Develop a comprehensive older adults screening tool for community dwelling older adults who attend congregate meal sites to assist in the evaluation of undernourishment or those at risk that is simple, faster, and less expensive

SUMMARY:
The COAST nutrition screening tool will be validated in 300 community-dwelling older adults in Florida.

DETAILED DESCRIPTION:
The population to be studied (n=300) will be individuals who are 60 years or older and participate in congregate meal sites or other community groups in Florida. Demographic information will be collected and participants will be assessed by the MNA® (Mini Nutrition Assessment) and screened by the COAST nutrition screening tool. Participants' hand grip strength and performance on the five times Sit to Stand test will be used to evaluate their functional status. Weight, height, mid-arm circumference and calf circumference will be measured as part of the MNA screening tool.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults 60 years and older.

Exclusion Criteria:

* Non-English speaking/reading

Ages: 60 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Older adults who attend congregate meal sites and other community groups in Florida will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
At Risk of Malnutrition | 1 year
  Number of subjects with an MNA® score of < 23.5

SECONDARY OUTCOMES:
Handgrip strength | 1 year
  Number of subjects with clinical weakness (<16 kg women; <26 kg men)
COAST | 1 year
  Association of COAST score to MNA® at risk of malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No